CLINICAL TRIAL: NCT01709955
Title: The Effects of Glucomannan on Weight Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northeast College of Health Sciences (Other)
Responsible Party: Principal Investigator, Denise Holtzman MS DC, Associate professor, Northeast College of Health Sciences
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-13
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Glucomannan
MeSH Terms: conditions — Obesity; Overweight | interventions — (1-6)-alpha-glucomannan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gucomannan (Experimental)
  Interventions: Dietary Supplement: Glucomannan
- Placebo pill (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Glucomannan — 750 MG of Glucomannan in capsule form
  Arms: Gucomannan
Other: Placebo — 750 mg of Cellulose powder in a capsule form
  Arms: Placebo pill

SUMMARY:
The purpose of this study is to determine if the herb, Glucomannan, is an effective non-pharmacological appetite suppressant for overweight or Class I obese patients. The study design will not include any other lifestyle changes which enhance weight loss in order to completely isolate the effects of Glucomannan as a non-pharmacological appetite suppressant.

ELIGIBILITY:
Inclusion Criteria:Subjects will be recruited based upon the category of them wanting to lose 50 pounds.

Subjects must be able to swallow the capsule whole with water.

Exclusion Criteria:

1. Self-reported use of prescription medication other than hormonal birth control (such as medication for diabetes, hypertension hypothyroidism, heart disease, cancer, etc.)
2. Pregnancy
3. Age younger than 21 or older than 60 years of age.
4. Screening for hypertension during the first laboratory visit that reveals a systole greater than 120 and a diastole greater than 90.
5. BMI calculations based upon height and weight measurements at the first laboratory visit that reveal a BMI less than 25 or greater than 35.
6. Self-reported iron-deficiency anemia, osteoporosis, and hypoglycemia.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 30 Days